CLINICAL TRIAL: NCT02872259
Title: A Phase Ib/II Randomised Open Label Study of BGB324 in Combination With Pembrolizumab or Dabrafenib/Trametinib Compared to Pembrolizumab or Dabrafenib/Trametinib Alone, in Patients With Advanced Non-resectable (Stage IIIc) or Metastatic (Stage IV) Melanoma
Brief Title: BGB324 in Combination With Pembrolizumab or Dabrafenib/Trametinib in Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Collaborators: BerGenBio ASA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015/1155
Record Dates: First submitted 2016-06-28; First posted 2016-08-19 (Estimated); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Melanoma
Keywords: metastatic melanoma; advanced Non-resectable melanoma
MeSH Terms: conditions — Melanoma | interventions — pembrolizumab; trametinib; dabrafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- BGB324 + pembrolizumab (Experimental): BGB324 capsules, 200 mg once daily + pembrolizumab 2 mg/kg IV every 3. week
  Treatment until disease progression, or unacceptable toxicity
  Interventions: Drug: BGB324+pembrolizumab
- BGB324 + dabrafenib and trametinib (Experimental): BGB324 capsules: Dose finding part of the study will determine if 100 mg once daily should be used for main part of the study or if 200 mg once daily once daily should be used.
  Dabrafenib capsules: 150 mg twice daily Trametinib tablets: 2 mg once daily
  Treatment until disease progression, or unacceptable toxicity
  Interventions: Drug: BGB324+dabrafenib and trametinib
- pembrolizumab (Active Comparator): Pembrolizumab 2 mg/kg IV every 3. week
  Treatment until disease progression, or unacceptable toxicity
  Interventions: Drug: pembrolizumab
- dabrafenib and trametinib (Active Comparator): Dabrafenib capsules:150 mg twice daily Trametinib tablets: 2 mg once daily
  Treatment until disease progression, or unacceptable toxicity
  Interventions: Drug: dabrafenib and trametinib

INTERVENTIONS:
Drug: BGB324+pembrolizumab — Combination
  Other Names: Keytruda
  Arms: BGB324 + pembrolizumab
Drug: BGB324+dabrafenib and trametinib — Combination
  Other Names: Tafinlar; Mekinist
  Arms: BGB324 + dabrafenib and trametinib
Drug: pembrolizumab — Monotherapy
  Other Names: Keytruda
  Arms: pembrolizumab
Drug: dabrafenib and trametinib — Combination
  Other Names: Tafinlar; Mekinist
  Arms: dabrafenib and trametinib

SUMMARY:
The purpose of the study is to assess the safety and efficacy of BGB324 given together with standard treatment, pembrolizumab or dabrafenib and trametinib, compared to standard treatment alone,

DETAILED DESCRIPTION:
This is an investigator initiated randomized randomized clinical phase 1b/2 clinical trial comparing safety and efficacy of the Axl inhibitor BGB324 in combination with pembrolizumab or dabrafenib+trametinib with that of pembrolizumab or dabrafenib+trametinib alone. Patients with non-resectable stage III or stage IV melanoma will be stratified based on BRAF mutation and tumor load to start dabrafenib+trametinib (BRAF mutation and high tumor load) or pembrolizumab (BRAF wild type or BRAF mutation and low tumor load) in first line. The patients will be randomized 2:1 to receive BGB324 in combination with pembrolizumab or dabrafenib+trametinib or to receive pembrolizumab or dabrafenib+trametinib alone. A 3+3 dose escalation will be performed for the combination of BGB324 and dabrafenib+trametinib. There is a major focus on predictive markers of treatment response evaluated in blood samples and biopsies.

ELIGIBILITY:
Inclusion Criteria:

1. Patients able to understand and willing to sign a written protocol specific informed consent and 18 years or older at the time of consent
2. Histologically confirmed advanced cutaneous melanoma that is either non-resectable (Stage IIIc) or metastatic (Stage IV) with:

   1. At least one measurable lesion as defined by RECIST 1.1 on CT or MRI scan and
   2. Documented progression of ≥1 measurable lesion
3. ECOG score 0 to 2 at screening
4. Availability of fresh or archival tumour tissue sample suitable for evaluation of predictive biomarkers of response
5. Male patients with female partners of childbearing potential and female patients of childbearing potential willing to practice highly effective birth control from screening, throughout the study and for at least 3 months following the last dose of study treatment (and if female of childbearing potential, has a negative serum pregnancy test in the 7 days before the first dose of study treatment)

Exclusion Criteria:

1. Prior first line systemic treatment for the treatment of Stage IIIb or Stage IIIc melanoma, including BRAF or MEK inhibitor (adjuvant immunomodulating agent treatment more than 6 months prior to first dose of study treatment is allowed)
2. Symptomatic central nervous system metastatic lesions as determined by the Investigator (patients with radiographically stable, asymptomatic lesions previously irradiated or surgically resected are eligible provided there is no need for systemic corticosteroids and treatment was completed at least 4 weeks before the first dose of study treatment)
3. History of malignancy other than melanoma within the last 2 years (basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix; isolated elevation in prostate specific antigen in the absence of histological or radiographic evidence of prostate cancer is allowed)
4. History of or current active autoimmune diseases, including but not limited to inflammatory bowel diseases, rheumatoid arthritis, autoimmune thyroiditis, autoimmune hepatitis, systemic sclerosis (scleroderma and variants), systemic lupus erythematosus, autoimmune vasculitis, autoimmune neuropathies (e.g. Guillain-Barré syndrome). Patients with vitiligo, or other non-serious autoimmune diseases based on the Investigator's assessment, are NOT excluded
5. ONLY FOR BRAF POSITIVE PATIENTS: History of retinal vein occlusion (RVO) or ongoing retinal pigment epithelial detachment (RPED)
6. History of the following cardiac conditions:

   1. Congestive cardiac failure of >Grade 2 severity (see Appendix 1) according to the New York Heart Association (defined as symptomatic at less than ordinary levels of activity)
   2. Ischemic cardiac event including myocardial infarction within 3 months prior to first dose of study treatment
   3. Uncontrolled cardiac disease, including unstable angina, uncontrolled hypertension (i.e. sustained systolic blood pressure >160 mmHg or diastolic blood pressure >90 mmHg), or need to change medication within 6 weeks of provision of consent due to lack of disease control
   4. History or presence of sustained bradycardia (≤55 bpm), left bundle branch block, cardiac pacemaker or ventricular arrhythmia. Note: Patients with a supraventricular arrhythmia requiring medical treatment, but with a normal ventricular rate are eligible
   5. Family history of long QTc syndrome; personal history of long QTc syndrome or previous drug-induced QTc prolongation
7. Known abnormal left ventricular ejection fraction on echocardiography or Multi Gated Acquisition (MUGA) scan (less than the lower limit of normal for a patient of that age at the treating institution or <45%, whichever is lower)
8. Current treatment with any agent known to cause Torsade de Points which cannot be discontinued at least five half-lives or two weeks prior to the first dose of study treatment
9. Screening 12-lead ECG with a measurable QTc interval calculated according to Fridericia's correction (QTcF) >450 ms
10. Inadequate organ function as defined by the following laboratory values:

    1. Haematological: absolute neutrophil count ≤1.5 x 109/L, platelets ≤100 x 109/L, haemoglobin ≤9.0 g/dL
    2. Renal: serum creatinine ≥1.5 x institutional upper limit of normal (ULN) and creatinine clearance ≥50 mL/minute
    3. Hepatic: total bilirubin ≥1.5 x institutional ULN, alanine transaminase (ALT) and aspartate transaminase (AST) ≥2.5 x institutional ULN or ≥5.0 x institutional ULN if liver metastases are present
    4. Coagulation: international normalised ratio or prothrombin time and activated partial thromboplastin time ≥1.5 x institutional ULN if not using anticoagulants (if patient is receiving anticoagulant therapy value must be within therapeutic range for the condition being treated)
11. Ongoing infection requiring systemic treatment. Patients who are on prophylactic anti infectives or who have been afebrile for 48 hours following the initiation of treatment are eligible
12. Known active infection with human immunodeficiency virus (HIV), hepatitis B or C viruses (screening not required)

    * Patients who have a history of hepatitis B infection are eligible provided they are hepatitis B surface antigen negative
    * Patients who have a history of hepatitis C infection are eligible provided they have no evidence of hepatitis C ribonucleic acid using a quantitative polymerase chain reaction assay at least 6 months after completing treatment for hepatitis C infection
13. Any conditions which may have significant impact on absorption of BGB324 or dabrafenib or trametinib from the gastrointestinal tract (including but not limited to, celiac disease or Crohn's disease, gastric or bowel resection)
14. Any severe or uncontrolled medical conditions which may jeopardise patient safety, compliance with the protocol, or interpretation of study results in the opinion of the Investigator
15. Current or recent (within last year) systemic treatment with immunosuppressive or immunomodulating agents (including systemic steroids intended for immunosuppressive effect), or other medications known to have significant impact on the immune system. Topical agents and inhaled steroids are permitted
16. Treatment with any medication with a narrow therapeutic index which is predominantly metabolised by cytochrome P450 (CYP)3A4 and cannot be stopped before the first dose of study treatment
17. Known hypersensitivity to pembrolizumab or BGB324 or excipients (including lactose intolerance)
18. ONLY FOR BRAF POSITIVE PATIENTS: Known hypersensitivity to dabrafenib or trametinib (including lactose intolerance)
19. Treatment with histamine receptor 2 inhibitors, proton pump inhibitors or antacids in the 7 days before the first dose of study treatment
20. Treatment with more than 40 mg prednisolone (or equivalent dose of systemic corticosteroid) which cannot be discontinued up to one week prior to starting BGB324. During the study this exclusion criteria is only applicable for patients receiving BGB324.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2017-02-13 (Actual); Primary Completion 2024-05-23 (Actual); Study Completion 2024-05-23 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) assessed according to RECIST Version 1.1 | through study completion, an average of 1 year
Number of participants with treatment-related adverse events as assessed by CTCAE v4.0 | through study completion, an average of 1 year

SECONDARY OUTCOMES:
Progression Free Survival (PFS) | ongoing evaluation, assessed up to 5 years
  From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 5 years
Duration of response | ongoing evaluation, an average of 1 year
  through study completion, an average of 1 year
Overall Survival (OS) | ongoing evaluation, an average of 2 year
  through study completion, an average of 2 year

CONTACTS AND LOCATIONS:
Overall Officials: Oddbjørn Straume, MD PhD, Principal Investigator — Haukeland University Hospital, 5021 Bergen, Norway
Locations (5):
- Norway (5):
  - Haukeland University Hospital, Bergen
  - Akershus Univerisity Hospital, Lørenskog
  - Oslo University Hospital, Radiumhospitalet, Oslo
  - University Hospital of North Norway, Tromsø
  - St. Olavs Hospital, Trondheim

IPD SHARING:
Plan to Share IPD: Undecided